CLINICAL TRIAL: NCT07072338
Title: PROMISE: Promoting Mental and Cognitive Health in Old Age Through Scalable Evidence-Based Interventions - Study Protocol for a Randomized Controlled Trial
Brief Title: Promoting Mental and Cognitive Health in Old Age Through Scalable Evidence-based Interventions
Acronym: PROMISE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Geneva, Switzerland (Other)
Responsible Party: Principal Investigator, Melanie Mack, Postdoctoral researcher at the Center for the Interdisciplinary Study of Gerontology and Vulnerabilities (CIGEV), University of Geneva, under the supervision of Professor Matthias Kliegel, University of Geneva, Switzerland
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 101080323
Record Dates: First submitted 2025-06-13; First posted 2025-07-18 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Well-Being, Psychological; Cognition; Ageing
Keywords: well-being; mental health; cognitive health; healthy aging; cognitive function; stress-management training; Acceptance and commitment therapy; cognitive training; lifrstyle intervention
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Stress management training Self-Help+ (SH+) (Experimental)
  Interventions: Behavioral: Stress management training
- Multodomain cognitive training (COG) (Experimental)
  Interventions: Behavioral: Multidomain cognitive training
- SH+ and COG combined (Experimental)
  Interventions: Behavioral: Stress management training; Behavioral: Multidomain cognitive training
- Podcast discussions (Active Comparator)
  Interventions: Behavioral: Social activities

INTERVENTIONS:
Behavioral: Stress management training — The stress management training is the WHO SH+ (Self-Help Plus) program, a low-intensity, group-based intervention developed by the World Health Organization to improve stress management and psychological flexibility. It combines pre-recorded audio sessions with an illustrated self-help guide and is based on Acceptance and Commitment Therapy (ACT). The program is delivered over five sessions and supported by a digital platform for at-home practice.
  Arms: SH+ and COG combined; Stress management training Self-Help+ (SH+)
Behavioral: Multidomain cognitive training — The multidomain cognitive training is a low-intensity, group-based intervention aimed at sustainably improving a healthy lifestyle, which in turn supports brain health and cognitive functioning. It combines pre-recorded audio sessions with an illustrated self-help guide and provides knowledge about aging and how to enhance three key lifestyle factors-social engagement, physical activity, and cognitive stimulation. The training uses metacognitive strategies and monitoring tools to help participants sustainably integrate these behaviors into their daily lives. The program is delivered over five sessions and supported by a digital platform for at-home practice.
  Arms: Multodomain cognitive training (COG); SH+ and COG combined
Behavioral: Social activities — The social activity intervention consists of a podcast discussion group in which participants listen to short podcasts on aging-related topics during each group session. Topics include driving (Session 1), intergenerational relationships (Session 2), technology (Session 3), the transition to retirement (Session 4), and travel (Session 5). These themes are deliberately chosen to be neutral and are not directly related to the techniques or content used to enhance well-being or cognitive functioning in the SH+ or COG interventions. The program is delivered over five sessions.
  Arms: Podcast discussions

SUMMARY:
Mental and cognitive health are key determinants of healthy and successful aging. These two domains are closely intertwined: while chronic stress can impair cognitive functioning, cognitive decline may in turn heighten stress and reduce overall well-being in older adults. This project aims to evaluate the effectiveness and scalability of a multidomain intervention to support mental and cognitive health in older adults. A single-blind, randomized, controlled 2×2 factorial trial will be conducted with a large sample of community-dwelling adults aged 65 years and older in the German- and French-speaking regions of Switzerland. Participants will be randomly assigned to one of four intervention arms: (1) WHO Self-Help Plus stress management training (SH+), (2) multidomain cognitive training focused on lifestyle and behavior change (COG), (3) a combined SH+ and COG intervention (SH+/COG), or (4) an active control group (CG) involving podcast listening and discussion. All interventions will include in-person group sessions, while the SH+, COG, and SH+/COG arms additionally offer a digital platform for self-guided home training. Primary outcomes (mental and cognitive health), secondary outcomes and moderators (cognitive functioning, stigma, self-efficacy, self-concept, loneliness, digital literacy, cognitive reserve, sociodemographic variables) will be assessed at baseline, post-intervention (10 weeks), and at 2- and 6-month follow-ups through a self-administered ambulatory assessment.

ELIGIBILITY:
Inclusion Criteria:

* Aged 65 years or older.
* Ability to speak and read the official language of their place of residence (French or German).
* Ability to use and access a digital device for a digital training platform provided for the training.

Exclusion Criteria:

* Aged below 65.
* Inability to use and lack of access to a digital device required for using the digital training platform.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Health related quality of life | Assessed before the intervention begins (pretest), after it concludes (10 weeks, posttest), and at two follow-ups: one at 2 months and another at 6 months post-intervention.
  Measurement tool: EuroQol Five-Dimensional Five-Level Scale (EQ-5D-5L; Herdman et al., 2011); Unit of measure: EQ-5D-5L index score (country-specific value set; range: -0.661 to 1.000 for Germany). Higher values on the EQ-5D index indicate better health status.
Well-being | Assessed before the intervention begins (pretest), after it concludes (10 weeks, posttest), and at two follow-ups: one at 2 months and another at 6 months post-intervention.
  Measurement tool: Capability Index for Older People, Scale (ICECAP-O; Gustafsson & Horder, 2022; Coast et al., 2008); Unit of measure: The ICECAP-O assesses five core dimensions of well-being relevant to older adults (attachment, security, role, enjoyment, control). ICECAP-O scores on the five core dimensions range from 1 to 4, with 1 being the lowest and 4 being the highest. These raw scores are then converted to tariff scores, ranging from 0 (representing absence of capability) to 1 (representing full capability).
Psychological distress | Assessed before the intervention begins (pretest), after it concludes (10 weeks, posttest), and at two follow-ups: one at 2 months and another at 6 months post-intervention.
  Measurement tool: Kessler Psychological Distress Scale (K6; Kessler et al., 2002); Unit of measure: K6 total score ranges from 0 to 24, with higher values indicating greater psychological distress.
Depression | Assessed before the intervention begins (pretest), after it concludes (10 weeks, posttest), and at two follow-ups: one at 2 months and another at 6 months post-intervention.
  Measurement tool: Geriatric Depression Scale - Short Form, Scale (GDS-SF; Sheikh & Yesavage, 1986); Unit of measure: GDS-SF total score ranges from 0 to 15, with higher scores indicating higher levels of depression.
Anxiety | Assessed before the intervention begins (pretest), after it concludes (10 weeks, posttest), and at two follow-ups: one at 2 months and another at 6 months post-intervention.
  Measurement tool: Geriatric Anxiety Inventory - Short Form, Scale (GAI-SF; Byrne & Pachana, 2010); Unit of measure: The GAI-SF total score ranges between 0 to 5, with higher scores representing higher anxiety levels.
Cognitive health | Assessed before the intervention begins (pretest), after it concludes (10 weeks, posttest), and at two follow-ups: one at 2 months and another at 6 months post-intervention.
  Measurement tool: Brain Care Score, Scale (self-designed scale based on Singh et al., 2023; Livingston et al., 2020; Ngandu et al., 2015); The Brain Care Score assesses six key dimensions known to be related to brain health: exercise, cognitive stimulation, social engagement, stress, sleep, and nutrition. Scores on the six dimensions range from 1 to 5. The total score ranges from 6 to 30, with higher scores indicating a lifestyle more supportive of brain health.
Health related quality of life | Assessed before the intervention begins (pretest), after it concludes (10 weeks, posttest), and at two follow-ups: one at 2 months and another at 6 months post-intervention.
  Measurement tool: EuroQol Five-Dimensional Five-Level Scale (EQ-5D-5L; Herdman et al., 2011); Unit of measure: EQ-5D-5L index score (country-specific value set; range: -0.661 to 1.000 for Germany) and Visual Analog Scale (VAS; range: 0-100). Higher values on the EQ-5D index indicate better health status, and higher values on the VAS also indicate better perceived health.

SECONDARY OUTCOMES:
Perceived health | Assessed before the intervention begins (pretest), after it concludes (10 weeks, posttest), and at two follow-ups: one at 2 months and another at 6 months post-intervention.
  Measurement tool: EuroQol Five-Dimensional Five-Level Scale (EQ-5D-5L; Herdman et al., 2011); Unit of measure: Visual Analog Scale (VAS; range: 0-100). Higher values on the VAS indicate better perceived health.

OTHER OUTCOMES:
Overall cognitive functioning | Assessed before the intervention begins (pretest), after it concludes (10 weeks, posttest), and at two follow-ups: one at 2 months and another at 6 months post-intervention.
  Measurement tool: Cognitive Telephone Screening Instrument, Scale (COGTEL, online version: E-COGTEL; Kliegel et al., 2007); Unit of measure: The total COGTEL score is derived from the sum of the weighted scores of each of the six subtests. A high score indicates better global cognitive functioning.
Abstract reasoning and fluid intelligence | Assessed before the intervention begins (pretest), after it concludes (10 weeks, posttest), and at two follow-ups: one at 2 months and another at 6 months post-intervention.
  Measurement tool: Raven Advanced Progressive Matrices - Short Form, Scale (APM; Arthur & Day, 1994; Raven et al., 1985); Unit of measure: The APM total score ranges from 0 to 12 points, with higher scores indicating a higher general cognitive ability.
Subjective cognitive complaints | Assessed before the intervention begins (pretest), after it concludes (10 weeks, posttest), and at two follow-ups: one at 2 months and another at 6 months post-intervention.
  Measurement tool: Subjective Cognitive Complaints Questionnaire (self-designed; Geerlings et al., 1999; Jessen, 2010; EIlis et al., 2014); Unit of measure: This instrument consists of five yes/no items that assess both perceived memory decline and related concerns.
Perceived age discrimination | Assessed before the intervention begins (pretest), after it concludes (10 weeks, posttest), and at two follow-ups: one at 2 months and another at 6 months post-intervention.
  Measurement tool: Perceived Experiences of Age Discrimination Scale (PAD; De Paula Couto et al., 2023); Unit of measure: The PAD total score ranges from 0 to 4, with higher scores indicating a greater frequency or intensity of perceived age discrimination.
Age-related stereotype threat | Assessed before the intervention begins (pretest), after it concludes (10 weeks, posttest), and at two follow-ups: one at 2 months and another at 6 months post-intervention.
  Measurement tool: Age-related Stereotype Threat Scale (not yet published version); Unit of measure: Higher total scores indicate greater age-related stereotype threat.
Self-efficacy | Assessed before the intervention begins (pretest), after it concludes (10 weeks, posttest), and at two follow-ups: one at 2 months and another at 6 months post-intervention.
  Measurement tool: Generalized Self-Efficacy Scale (GSE; Jerusalem & Schwarzer, 1992); Unit of measure: The total GSE score ranges from 10 to 40, with higher values indicating a stronger generalized sense of self-efficacy.
Self-concept | Assessed before the intervention begins (pretest), after it concludes (10 weeks, posttest), and at two follow-ups: one at 2 months and another at 6 months post-intervention.
  Measurement tool: Subjective Aging Perception Scale (SAPS; De Gracia et al., 1999); Unit of measure: The SAPS assesses four dimensions of individuals' perceptions and attitudes toward their own aging process (perceived self-care, perceived social resources, cognitive self-competence, perceived time structure). Scores on the four dimensions vary between 3 and 20, with higher scores indicating more positive perceptions of aging.
Social support | Assessed before the intervention begins (pretest), after it concludes (10 weeks, posttest), and at two follow-ups: one at 2 months and another at 6 months post-intervention.
  Measurement tool: Lubben Social Network Scale - 6 items (LSNS-6; Lubben et al., 2006); Unit of measure: The total LSNS-6 score ranges from 0 to 30. Higher scores indicate a larger, more active social network and stronger social connections.
Loneliness | Assessed before the intervention begins (pretest), after it concludes (10 weeks, posttest), and at two follow-ups: one at 2 months and another at 6 months post-intervention.
  Measurement tool: De Jong Gierveld 6-item Loneliness Scale (DJGLS-6; De Jong Gierveld & Van Tilburg, 2006); Unit of measure: The DJGLS-6 total score ranges from 1 to 5, with higher scores indicating greater loneliness.
Digital literacy | Assessed before the intervention begins (pretest).
  Measurement tool: Senior Technology Acceptance Model - Short Form, Scale (Short STAM; Chen & Lou, 2020); Unit of measure: The Short STAM total score ranges from 14 to 140, with higher scores indicating greater technology acceptance.
Cognitive reserve | Assessed before the intervention begins (pretest).
  Measurement tool: Cognitive Reserve Index questionnaire, Scale (CRIq; Nucci et al., 2012); Unit of measure: The total CRIq score is standardized: the average is 100, with a standard deviation of 15. Higher values indicate greater cognitive reserve.
Subjective social status | Assessed before the intervention begins (pretest).
  Measurement tool: MacArthur Scale of Subjective Social Status, Scale (MacArthur SSS Scale; Adler et al., 2000); Unit of measure: The MacArthur SSS score ranges from 1 to 100, with higher values indicating a higher perceived social status.
Cost of services | Assessed before the intervention begins (pretest), after it concludes (10 weeks, posttest), and at two follow-ups: one at 2 months and another at 6 months post-intervention.
  Measurement tool: Client Service Receipt Inventory (CSRI; Chisholm et al., 2000); Unit of measure: Different questions gather information on health and social care service use, informal care, employment and income, living situation and housing, as well as medication and treatment adherence. This information will be used to estimate total costs per participant over the past two months.
Session attendance | Between pretest and posttest (10 weeks).
  Measurement tool: Facilitator Attendance Logs; Unit of measure: Number of attended sessions: ranges from 0 to 10, with higher numbers indicating greater session attendance.
Usage of digital platform | From pretest until follow-up 2 (8 months).
  Measurement tool: Digital platform usage data; Unit of measure: The platform gathers information on different usage markers such as number of logins, number of completed training sessions, total time spent on the platform, and number of days with at least one activity. Higher values indicate greater engagement with the digital intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Center for the Interdisciplinary Study of Gerontology and Vulnerabilities, Geneva, Canton of Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Project website — https://advancementalhealth.ku.dk/activities/older-adults/
- See also: Information for participants — https://cigev.unige.ch/advance